CLINICAL TRIAL: NCT03315364
Title: A Multinational, Multicenter, Open-label, Phase II/III Clinical Trial to Evaluate the Efficacy and Safety of Liporaxel® (Oral Paclitaxel) Compared to Taxol® (IV Paclitaxel) as First-line Therapy in Patients With Recurrent or Metastatic HER2 Negative Breast Cancer
Brief Title: Oral Paclitaxel Trial In Recurrent and Metastatic Breast Cancer As 1st Line Therapy
Acronym: OPTIMAL
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107CS-5
Record Dates: First submitted 2017-09-28; First posted 2017-10-20 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Recurrent or Metastatic Breast Cancer
Keywords: Recurrent breast cancer; Metastatic breast cancer; MBC; Firstline chemotherapy; Paclitaxel; Liporaxel; Taxol
MeSH Terms: conditions — Recurrence; Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: 1. Phase II clinical trial
     * Multicenter, Open-label, Single arm, Simon's optimal two-stage design
  2. Phase III clinical trial
     * Multicenter, Prospective Randomized Open-label Blinded Endpoint (PROBE) design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liporaxel® (oral paclitaxel) (Experimental): * 28 days (4 weeks) will be set as one cycle of administration and Liporaxel® will be administered for 3 weeks, twice a day, every morning and evening (D1, D8, D15) and will take a week off on 4th week.
  * Liproaxel® 200mg/m2 will be orally administered twice a day (morning, evening) 1 hour after meal for D1, D8, D15 of every cycle. 10 hour-interval is recommended for between each administration.
  Interventions: Drug: Oral paclitaxel
- Taxol® (IV paclitaxel) (Active Comparator): * 28 days (4 weeks) will be set as one cycle and for every 3 week administration, 1 week off dose period will be given.
  * Taxol® 80mg/m2 will be administered via IV and it must be diluted before drip administration. Dilute with 0.9% sodium chloride injection solution to make final concentration of 0.3-1.2 mg/mL.
  Interventions: Drug: Paclitaxel injection

INTERVENTIONS:
Drug: Oral paclitaxel — Oral administration on D1, D8 and D15 of 4-week cycle until progression, unacceptable toxicity or withdrawal of informed concent
  Other Names: Liporaxel®
  Arms: Liporaxel® (oral paclitaxel)
Drug: Paclitaxel injection — Premedication, intravenous infusion on D1, D8 and D15 of 4-week cycle until progression, unacceptable toxicity or withdrawal of informed concent
  Other Names: Taxol®
  Arms: Taxol® (IV paclitaxel)

SUMMARY:
To compare and evaluate the efficacy and safety of Liporaxel® solution (oral paclitaxel) and Taxol® (IV paclitaxel) on recurrent or metastatic breast cancer.

ELIGIBILITY:
Key inclusion/exclusion criteria

* Histologically or cytologically confirmed to have recurrent, or metastatic breast cancer.
* Measurable disease (revised RECIST, version 1.1).
* Hormone receptor (ER/PR) positive or negative, HER2 negative.
* Subjects were eligible for the study regardless of their previous lines of endocrine therapy.
* No prior chemotherapy is allowed in metastatic disease.
* Subjects who administrated the last dose of taxane class drug ≥12months ago as from the first administration day.
* ECOG performance status ≤1.
* Neuropathy grade <2.
* Subjects with central nervous system metastasis should be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
[Phase II] Objective Response Rate (ORR) | Participants will be followed every 6 weeks until progression, an expected average of 9 months.
  Objective Response Rate (ORR) is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (v.1.1) criteria.
[Phase III] Progression Free Survival (PFS) | From date of randomization, assessed up to 18 months.
  Progression Free Survival (PFS) is defined as the time from date of randomization until the date of first documented progression or death

SECONDARY OUTCOMES:
[Phase II] Progression Free Survival (PFS) | From date of randomization, assessed up to 18 months.
  Progression Free Survival (PFS) is defined as the time from date of randomization until the date of first documented progression or death
[Phase III] Objective Response Rate (ORR) | Participants will be followed every 6 weeks until progression, an expected average of 9 months.
  Objective Response Rate (ORR) is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (v.1.1) criteria.
[Phase II&III] Overall Survival(OS) | Until 6 months after the last participant is enrolled, assessed minimum to 18 months.
  Overall survival(OS) is defined as the time from the date of inclusion to the date of death, regardless of the cause of death.
[Phase II&III] Time to Treatment Failure(TTF) | through study completion, an expected average of 4.5 year.
  TTF is defined as the time from the randomization date to the date of discontinuation of treatment, regardless of the cause.
[Phase II&III] Disease Control Rate(DCR) | through study completion, an expected average of 4.5 year.
  DCR is defined as the percentage of subjects who were evaluated for complete response(CR), partial response(PR), and stable disease(SD) as the best response among from randomization to End of treatment(EOT).
[Phase II&III] Quality of life(QoL) | C1D1, C2D1, C4D1, C7D1, C10D1 (each cycle is 28 days) and study completion, up to 18 months.
  To evaluate changes versus baseline using the EQ-5D.
Incidence of Treatment-Emergent Adverse Events [Safety] | Up to 28 days after last investigational product administraion.
  Number and Description of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Sung-bae Kim, M.D., Ph.D, Principal Investigator — Asan Medical Center
Locations (51):
- Bulgaria (3):
  - Oncology Complex Center - Burgas'' Ltd., Medical Oncology Department, Burgas
  - Multi-profile Hospital for Active Treatment Uni Hospital Ltd. Medical Oncology Department, Panagyurishte
  - Medical Center Nadezhda Clinical" Ltd.,, Sofia
- China (18):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy Of Medical Sciences, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Hainan Medical College, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tianjin Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shangdong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong university, Xi’an, Shanxi
  - West China School Of Medicine Sichuan University, Chengdu, Sichuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang University School Of Medicine Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Hungary (2):
  - Tolna County Balassa János Hospital, Szekszárd
  - Szent Borbála Hospital, Tatabánya
- Serbia (7):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Clinical Hospital Center Bežanijska Kosa, Department of Oncology, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Health Center Kladovo, Oncology Department, Kladovo
  - Clinical Center Kragujevac Center of Oncology and Radiotherapy, Kragujevac
  - General Hospital Krusevac, Outpatient Clinic for chemotherapy, Kruševac
  - Clinical Center Niš, Clinic for Oncology, Niš
- South Korea (21):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Cha University Cha Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Gang Neung Asan Hospital, Gangneung
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Catholic University of Korea Seoul ST. Mary's Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Uijeongbu ST. Mary's Hospital, Uijeongbu-si

REFERENCES:
- [Derived] Kim SB, Seo JH, Ahn JH, Kim TY, Kang SY, Sohn J, Yang Y, Park KH, Moon YW, Lim S, Kang MJ, Yoon KE, Cho HJ, Lee KS. Phase II study of DHP107 (oral paclitaxel) in the first-line treatment of HER2-negative recurrent or metastatic breast cancer (OPTIMAL study). Ther Adv Med Oncol. 2021 Dec 15;13:17588359211061989. doi: 10.1177/17588359211061989. eCollection 2021. PMID 34925553